CLINICAL TRIAL: NCT04434755
Title: Wellness and Distress in Health Care Professionals Dealing With End of Life and Bioethical Issues (WeDistressHELL)
Brief Title: Wellness and Distress in Health Care Professionals Dealing With End of Life and Bioethical Issues
Acronym: WeStressHELL
Status: Completed | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: I.R.C.C.S. Fondazione Santa Lucia (Other); Istituto Clinico Humanitas (Other); University of Pavia (Other)
Responsible Party: Sponsor
Other Study IDs: ICS Maugeri CE 2211
Record Dates: First submitted 2020-06-08; First posted 2020-06-17 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2020-06

CONDITIONS: Burnout, Professional
Keywords: burnout; distress; wellness; end of life; bioethics
MeSH Terms: conditions — Burnout, Professional; Burnout, Psychological; Death

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- health care professionals in palliative care: health care professionals in palliative care
  Interventions: Other: health care professionals' exposure to bioethical issues
- health care professionals in neurorehabiliation: health care professionals in neurorehabiliation
  Interventions: Other: health care professionals' exposure to bioethical issues

INTERVENTIONS:
Other: health care professionals' exposure to bioethical issues — health care professionals were differentiated considering the work context and the type of patients cured

SUMMARY:
Burnout, fatigue, distress and negative issues are in health care providers with different percentages. To date, little is known about the experience of burnout, fatigue and distress related with end of life and bioethical issues.

The main aim of this study is to quantify burnout and identify a set of variables (meaning of life, stress, moral distress, ethical climate, resilience, positive and negative affects) that may impact on professionals dealing with end-of-life and bioethics issues in their working life.

The project is an observational multicentre cross-sectional study, population-based.

The target population is composed by psychologists, nurses and other healthcare providers dealing with end-of-life/palliative care and other conditions.

The study will be conducted using a mixed methods, using both quantitative and qualitative approaches.

Regarding the quantitative approaches, standardized questionnaires will be administered anonymously to each participant in one time only. Concerning the qualitative approaches, semi-structured interviews will be carried out until the saturation of categories is reached according to the Grounded Theory methodology It is mainly attended that this project may shed light on wellness and distress related to end-of-life and bioethical issues faced in working life by health care providers, considering not only risk factors but also protective and positive ones.

The quantitative part of the research is supposed to identify the dimension of burnout in this health-care professionals category and to better clarify the role of some variables (meaning of life, stress, moral distress, ethical climate, resilience, positive and negative affects) that may modulate and affect wellness and distress experienced by this category of workers.

The qualitative part of the study will help to frame better the issue, detecting the main demanding aspects.

DETAILED DESCRIPTION:
Burnout, fatigue, distress and negative issues are well known in health care providers with different percentages.

This issue is internationally considered relevant; physicians have 36% more probability of developing burnout with respect to the American high school graduated population and, in general, medical students, residents/fellows, and early career physicians are more likely to suffer from burnout compared to the general population. Moreover, between 2011 and 2014, the trend of job satisfaction and burnout was getting worse in these worker categories. This condition has to be seriously taken in consideration; indeed, chronic distress and burnout in health care providers affect both the quality of patient care and satisfaction, as well as the employee professional quality of life and psychological and physical wellbeing.

Risk factors are various and the most relevant include work features, interpersonal relationships and personal factors. However, only recently literature has focused on positive and protective factors which modulate too the relationship between the health care professional and her/his job. To date, little is known about the experience of burnout, fatigue and distress related with end of life and bioethical issues in everyday working life.

What emerges from qualitative studies is that a relevant source of distress is linked to the physicians and nurses' necessity to take bioethical decisions against their personal values, and another source of distress arises from balancing family, institutional and moral constraints.

According to quantitative researches, the exposure to death and dying results in distress, fatigue and impoverishment of professional quality of life. Moreover, a review reports that critical care nurses experience their most stressful job situation when they have to manage with the unnecessary prolongation of life of their patients on the bases of family's desire. Indeed, a risk factor to burnout seems to be the ethical decision-making regarding end of life and foregoing life-sustaining therapy. Another qualitative and quantitative review shows that health care practitioners' end-of-life decision making may contribute to the distress and burnout experience.

Contemporary medical practice implies an increasing amount of bioethical issues to manage and this fact may constrain physicians and health care professionals to experience relevant distressing and high demanding situations.

General objective The main aim of this study is to quantify burnout and identify a set of variables (meaning of life, stress, moral distress, ethical climate, resilience, positive and negative affects) that may impact on professionals dealing with end-of-life and bioethics issues in their working life by quantitative and qualitative methods.

Specific objectives - 1 to estimate the prevalence of the subjective perception of burnout among health-care professionals dealing with end-of-life and bioethical issues. 2: to evaluate possible relations among some influential variables (meaning of life, stress, moral distress, ethical climate, resilience, positive and negative affects) and burnout and wellness/distress among health-care professionals dealing with end-of-life and bioethical issues.

Methods Study design The project is an observational multicentre cross-sectional study, population-based.

Population The target population is composed by psychologists, nurses and other healthcare providers dealing with end-of-life/palliative care and other conditions possibly characterized by bioethical problems. Therefore, no sample size is needed.

All the healthcare professionals working in unit of end-of-life/palliative care and other conditions characterized by bioethical problems in three private Institutions (IRCCS): Istituti Clinici Scientifici Maugeri Spa SB, Humanitas Research Hospital - Rozzano (Milan) and I.R.C.C.S. Santa Lucia - Centro Riabilitativo - Roma (Roma) will be eligible and invited to participate at the study.

Since all the eligible will be enrolled the study is population based and no sample size is needed. Nevertheless achievement of at least 80% of responders will be fixed to ensure internal validity and minimizing selection bias.

There will be the possibility to extend the study in other countries too (to now ongoing contact with Croatia, Cyprus, Poland, Portugal) to maximize the generalizability of results.

Primary end point The subjective perception of burnout will be measured by Maslach Burnout Inventory - General Survey (MBI GS): a brief scale assessing the three dimensions of burnout: emotional exhaustion, depersonalization and professional efficacy.

Procedure The study will be conducted using a mixed methods, using both quantitative and qualitative approaches.

Regarding the quantitative approaches, standardized questionnaires will be administered anonymously to each participant in one time only. Only a numerical code will identify the participant's questionnaires battery. Participant's information linked to the numerical code will be encrypted and kept in security by a password. The access to this sensitive data will be possible only to authorised persons involved in the research.

Concerning the qualitative approaches, semi-structured interviews will be carried out until the saturation of categories is reached according to the Grounded Theory methodology.

The qualitative and quantitative part of the research will be carried out in Italy. Afterwards, the quantitative part only will be extended to other foreign countries interested to be involved in the research. These Institution will be further identified during the 13th World Conference on Bioethics, Medical Ethics & Health Law at the end of 2018 (Jerusalem, November 27th -29th, 2018). An amendment to research protocol will be presented if necessary.

Data collection will began according to previous agreements with the professionals and their Institution too.

Instruments

For the quantitative part of the study, the following instruments (Annex 3) will be used:

* MBI GS - Maslach Burnout Inventory - General Survey: a brief scale assessing the three dimensions of burnout: emotional exhaustion, depersonalization and professional efficacy;
* SMILE - Schedule for Meaning in Life Evaluation: a short open- and close-answer questionnaire assessing the individual meaning in life;
* MASI-R - Maugeri Stress Index: a brief questionnaire assessing work-related psychological stress;
* MDS-R - Moral Distress Scale-Revised: a brief scale scored by clinicians in terms of frequency and intensity assessing moral distress;
* HECS - Hospital Ethical Climate Survey: a short scale assessing ethical climate in the hospital perceived by healthcare professionals;
* CDS-RISC-10 - Connor-Davidson Resilience Scale: a 10 items questionnaire assessing resilience;
* PANAS - Positive Affect and Negative Affect Scale: a brief self-report measure assessing positive and negative dispositional dimensions.

Socio-demographic characteristics (i.e. sex, age, years of occupation in the unit) will be also collected.

For the qualitative part of the study, a semi-structured interview will be constructed according to literature suggestions on the same constructs assessed by the instruments cited above and on the bases of the Grounded Theory (GT) qualitative approach.

Statistical analysis Quantitative data will be summarized as mean with standard deviation, or median with 25th and 75th centile. Qualitative data will be described by percentages. Relationships between the scores will be described by the appropriate correlation coefficients. The appropriate bivariate analyses will be applied. The crude prevalence of subjective perception of burnout with the exact 95% confidence interval (95%CI) will be estimated. The association between the prevalence of burnout and the meaning of life, stress, moral distress, ethical climate, resilience, positive and negative affects will be investigated by logistic regression model and the effect of all these factors will be evaluated by Likelihood Ratio test.

Analyses for quantitative and qualitative data will be made using SPSS Statistics Standard (Statistics Standard - Statistical Package for Social Science (IBM Site). A p-value less than 0.05 will be considered significant.

The qualitative analysis of the semi-structured interviews will be carried out by means of the GT methodology, with the support of the open source R package for Qualitative Data Analysis (RQDA) purposely designed. This approach allows generating information thorough an iterative process involving continuous sampling and analysis of data derived from the concrete setting and, as a consequence, strongly "grounded" in the real experience

Study duration Even if the cross sectional design is planned, it will be necessary several time to conduct the interviews. So at least 12 months will be planned to develop the quantitative and qualitative approach.

Time Table -Time: first 18 months Recruitment of participants within the 2nd month.

From 3rd month to 14th month:

Quantitative part: administration of the standardized questionnaires, implementation of data in the database (data entry), and statistical analyses.

Qualitative part: semi-structured interviews data collection, transcriptions and analysis will be carried out in the same time and until the saturation of the emerged categories, according to the GT methodology

-Time: from 19th to 30th month

Expected results It is mainly attended that this project may shed light on wellness and distress related to end-of-life and bioethical issues faced in working life by health care providers, considering not only risk factors but also protective and positive ones according to the current international trend of research.

The quantitative part of the research is supposed to identify the dimension of burnout in this health-care professionals category and to better clarify the role of some variables (meaning of life, stress, moral distress, ethical climate, resilience, positive and negative affects) that may modulate and affect wellness and distress experienced by this category of workers.

The qualitative part of the study will help to frame better the issue, detecting the main demanding aspects in order to propose a grounded theory explaining the connections between wellness and distress related to end-of-life and bioethical issues in the working place.

Implications The implications may be of paramount relevance in the health care system. Indeed, worldwide advances in medical sciences and society transformations inevitably imply an ever-growing need of workers involved in palliative care and chronic disease units, as well as ever-proliferating bioethical quandaries impacting on the health care professionals' wellness.

From a theoretical point of view, these results could orientate the future research and enrich the growing amount of bioethical knowledge, in particular regarding aspects impacting on the quality of health care providers' working life.

From a practical point of view; implications may be:

* This study may help to focus on risk and protective factors to be monitored during the health care provider's career. The attended results may provide information useful for personal resources and for preventing distress experienced in daily medical practice dealing with end-of-life and bioethical issues.
* New insights on conditions of professionals who deal constantly with ever-increasing bioethical issues may provide suggestions on parameters, guidelines and legislation.
* These new insights may impact indirectly to the society since, "care of the patient requires care of the provider". Indeed, health care professionals' distress is a condition depleting the relationship with the patient and, as a consequence, also the quality and the adherence to the treatment besides to an unnecessary increase of care costs

ELIGIBILITY:
Inclusion Criteria:

psychologists, nurses and other healthcare providers dealing with end-of-life/palliative care and other conditions possibly characterized by bioethical problems.

Exclusion Criteria:

not signing the consent to participate to the study

-

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the healthcare professionals working in unit of end-of-life/palliative care and other conditions characterized by bioethical problems in three private Institutions (IRCCS): Istituti Clinici Scientifici Maugeri Spa SB, Humanitas Research Hospital - Rozzano (Milan) and I.R.C.C.S. Santa Lucia - Centro Riabilitativo - Roma (Roma) will be eligible and invited to participate at the study.
Sampling Method: Non-Probability Sample
Enrollment: 317 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
to estimate the prevalence of the subjective perception of burnout among health-care professionals dealing with end-of-life and bioethical issues. | 2018-2020
  Prevalence of the subjective perception of burnout among health-care professionals dealing with end-of-life and bioethcial issues

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Istituto Clinico Humanitas, Milan
  - Istituti Clinici Scientifici Maugeri IRCCS, Pavia
  - Fondazione Santa Lucia IRCCS, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hynes J, Maffoni M, Argentero P, Giorgi I, Giardini A. Palliative medicine physicians: doomed to burn? BMJ Support Palliat Care. 2019 Mar;9(1):45-46. doi: 10.1136/bmjspcare-2018-001731. No abstract available. PMID 30782969
- [Background] Maffoni M, Argentero P, Giorgi I, Hynes J, Giardini A. Healthcare professionals' moral distress in adult palliative care: a systematic review. BMJ Support Palliat Care. 2019 Sep;9(3):245-254. doi: 10.1136/bmjspcare-2018-001674. Epub 2019 Jan 12. PMID 30636204
- [Background] Zanatta F, Maffoni M, Giardini A. Resilience in palliative healthcare professionals: a systematic review. Support Care Cancer. 2020 Mar;28(3):971-978. doi: 10.1007/s00520-019-05194-1. Epub 2019 Dec 6. PMID 31811483
- [Background] Maffoni M, Argentero P, Giorgi I, Giardini A. Healthcare professionals' perceptions about the Italian law on advance directives. Nurs Ethics. 2020 May;27(3):796-808. doi: 10.1177/0969733019878831. Epub 2019 Oct 20. PMID 31631774
- [Background] Maffoni M, Argentero P, Giorgi I, Giardini A. Underneath the White Coat: Risk and Protective Factors for Palliative Care Providers in Their Daily Work. J Hosp Palliat Nurs. 2020 Apr;22(2):108-114. doi: 10.1097/NJH.0000000000000623. PMID 31977533
- [Background] Maffoni M, Sommovigo V, Giardini A, Paolucci S, Setti I. Dealing with ethical issues in rehabilitation medicine: The relationship between managerial support and emotional exhaustion is mediated by moral distress and enhanced by positive affectivity and resilience. J Nurs Manag. 2020 Jul;28(5):1114-1125. doi: 10.1111/jonm.13059. Epub 2020 Jun 23. PMID 32495373